CLINICAL TRIAL: NCT04559776
Title: Reliability and Sources of Variability of 3D Kinematics and Muscle Activation Analysis of Newly-acquired Gait in Toddlers With a Typical Development and a Unilateral Cerebral Palsy
Brief Title: Reliability of Newly-acquired Gait in Toddlers With a Typical Development and a Unilateral Cerebral Palsy
Acronym: ReliabBB-AQM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Clinical Center for Neuropsychomotor Recovery for Children Dr. Nicolae Robanescu (Other)
Collaborators: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 8463/2016
Record Dates: First submitted 2020-09-01; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Gait, Spastic; Reliability
Keywords: toddlers; 3D motion analysis; EMG; reliability
MeSH Terms: conditions — Gait Disorders, Neurologic | interventions — Gait Analysis

STUDY DESIGN:
Intervention Model Description: cross-sectional study with 2 groups of toddlers (with typical developing and with unilateral cerebral palsy) recorded twice in gait analysis within 30 days interval
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- typically developing toddlers (Experimental): toddlers with a typical development and with less than 3 years old and less than 6 months of independent walking
  Interventions: Other: gait analysis
- unilateral cerebral palsy toddlers (Experimental): toddlers with a unilateral cerebral plasy and with less than 3 years old and less than 6 months of independent walking
  Interventions: Other: gait analysis

INTERVENTIONS:
Other: gait analysis — gait analysis with 3D optoelectronic system and surface EMG

SUMMARY:
gait reliability study of toddlers with typically developing and with unilateral cerebral palsy during the first 6 months of independent walking

DETAILED DESCRIPTION:
This study aim to assess lower limb kinematics and muscle EMG reliability during gait in typically developing toddlers and in toddlers with unilateral cerebral palsy with less than 6 months of independent walking experience and secondary to determine three sources of variability (between subjects, between sessions and between trials) using an optoelectronic system and a surface EMG system. The third aim was to identify the most reliable gait parameters.

This was a cross-sectional study conducted between January 2016 and May 2018 in the Motion Analysis Laboratory of the National Rehabilitation Center for Children (NRCC) "Dr. N. Robanescu", Bucharest (Romania). The toddlers with UCP were recruited among the inpatients and outpatients of the Pediatric Rehabilitation department. TD toddlers were recruited among the siblings of the toddlers with UCP and the children of people known to the investigators. Given the exploratory nature of this study, the target size of each group was set to a minimum of 10 participants per group.Toddlers from both groups were younger than 3 years old and independent walking experience of maximum 6 months. Every child was proposed to be evaluated in two gait analysis sessions within a period of 30 days. The second gait analysis session was planned approximately at 14 days from the first one. The two sessions were performed by the same experienced assessor.

The toddlers walked barefoot at self-selected pace. Each toddler was equipped with 19 reflective markers and 8 surface EMG electrodes. Data was collected with a BTS motion capture system equipped with 8 infrared cameras and 8 channels EMG system. The biomechanical model used was "Helen Hayes with medial markers".The EMG electrodes were positioned according to the SENIAM recommendations over the rectus femoris, the medial hamstrings, the tibialis anterior and the triceps surae.Visual 3D software (C-motion, Rockville, MD, USA) was used to build the kinematic model and identify gait cycles. A qualitative analysis was conducted for each gait cycle and each child in order to exclude the cycles during running or non-straight walking. Data was filtered and normalized. Three sources of variability (between subjects, between sessions and between trials) for kinematics and EMG data were quantified by calculating the standard deviations for each source.Standard Error of Measurement (SEM) for intertrials and intersessions were also calculated. For TD toddlers, a single value was reported as the quadratic mean for the right and left sides.

ELIGIBILITY:
Inclusion Criteria:

Toddlers from both groups were included in this study if they met the following inclusion criteria:

* up to 3 years of age,
* maximum independent walking experience of 6 months, and
* able to walk 5 metres without falling and with no technical assistance. Regarding the UCP group, one additional inclusion criterion was added: right or left hemiparesis with a typical history of CP (prematurity, before birth stroke, acute foetal distress/ birth hypoxia, brain malformations...).

Regarding the TD group, two additional inclusion criteria were: typical development and independent gait acquired before the age of 18 months.

-

Exclusion Criteria:

Toddlers from both groups were excluded in case of

* trauma to the lower limbs in the last 6 months,
* a known skin allergy to any adhesive product, and
* any lower limb surgery. Toddlers in the UCP group were also excluded if they had botulinum toxin injections in the lower limb muscles in the previous 3 months.

Toddlers in the TD group were also excluded in the presence of a known neurological and/ or orthopaedic disorder.

Ages: 10 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
intertrials and intersessions kinematic reliability | 3 years
  Assess lower limb joint angles reliability during gait in TD toddlers and with toddlers with unilateral cerebral palsy (UCP) with less than 6 months of independent walking experience by calculating the Standard Error of Measurement (SEM) for each joint of the lower limb and each motion plane and in each group of toddlers (TD and UCP). For UCP toddlers, the SEM was calculated separately for the affected and the non-affected sides. SEM values for joint angles are expressed in degrees.
intertrials and intersessions EMG reliability | 3 years
  Assess lower limb reliability of the muscular EMG envelops during gait in TD toddlers and with toddlers with unilateral cerebral palsy (UCP) with less than 6 months of independent walking experience by calculating the Standard Error of Measurement (SEM) for of the four muscles studied (rectus femoris, medial hamstrings, tibialis anterior and triceps surae) and in each group of toddlers (TD and UCP). For UCP toddlers, the SEM was calculated separately for the affected and the non-affected sides. SEM values for EMG envelopes have no units of measure since the EMG envelope of a muscle is normalized by the maximum amplitude of the EMG signal of that muscle for all gait cycles for a subject.

SECONDARY OUTCOMES:
sources of variability for kinematics | 3 years
  Assess 3 sources of gait variability (intersubjects, intersessions, intertrials) during gait in TD toddlers and with toddlers with unilateral cerebral palsy (UCP) with less than 6 months of independent walking experience, by calculating the Standard Deviation (SD) for each joint and each motion plane of lower limb joint and in each group of toddlers (TD and UCP). For UCP toddlers, the SD was calculated separately for the affected and the non-affected sides. SD values for joint angles are expressed in degrees.
sources of variability for EMG | 3 years
  Assess 3 sources of gait variability (intersubjects, intersessions, intertrials) of the muscular EMG envelops during gait in TD toddlers and with toddlers with unilateral cerebral palsy (UCP) with less than 6 months of independent walking experience by calculating the Standard Deviation (SD) for of the four muscles studied (rectus femoris, medial hamstrings, tibialis anterior and triceps surae) and in each group of toddlers (TD and UCP). For UCP toddlers, the SD was calculated separately for the affected and the non-affected sides. SD values for EMG envelopes have no units of measure since the EMG envelope of a muscle is normalized by the maximum amplitude of the EMG signal of that muscle for all gait cycles for a subject.

OTHER OUTCOMES:
identify the most reliable kinematic parameters | 3 years
  identify those joints and planes where the Standard Error of Measurement (SEM) calculated for primary outcome have values below 5 degrees.

IPD SHARING:
Plan to Share IPD: No